M16-011 – Statistical Analysis Plan Version 6.0 – 23 November 2020

# **Statistical Analysis Plan for Study M16-011**

A Phase 3, Randomized, Double-Blind Study Comparing Risankizumab to Placebo in Subjects with Active Psoriatic Arthritis (PsA) Who Have a History of Inadequate Response to or Intolerance to at Least One Disease Modifying Anti-Rheumatic Drug (DMARD) Therapy

Date: 23 November 2020

Version 6.0

# **Table of Contents**

| 1.0 | Introduction | 6 |
|---|---|---|
| 2.0 | Study Design and Objectives | 6 |
| 2.1 | Objectives | 6 |
| 2.2 | Study Design Overview | 7 |
| 2.3 | Treatment Assignment and Blinding | 9 |
| 2.4 | Sample Size Determination | 9 |
| 3.0 | Endpoints | 9 |
| 3.1 | Primary Endpoint(s) | 9 |
| 3.2 | Secondary Endpoint(s) | 9 |
| 3.3 | Additional Efficacy Endpoints | 11 |
| 3.4 | Safety Endpoints | 14 |
| 3.5 | Additional Endpoints | 14 |
| 4.0 | Analysis Populations | 14 |
| 5.0 | Subject Disposition | 14 |
| 6.0 | Study Drug Duration and Compliance | 15 |
| 7.0 | Demographics, Baseline Characteristics, Medical | |
| | History, and Prior/Concomitant Medications | |
| 7.1 | Demographics and Baseline Characteristics | 16 |
| 7.2 | Medical History | 19 |
| 7.3 | Prior and Concomitant Medications | 20 |
| 8.0 | Efficacy Analyses | 20 |
| 8.1 | General Considerations | 20 |
| 8.2 | Handling of Missing Data and Intercurrent Events | 22 |
| 8.3 | Primary Efficacy Endpoint and Analysis | 25 |
| 8.3.1 | Primary Efficacy Endpoint | 25 |
| 8.3.2 | Handling of Missing Data and Intercurrent Event for the Primary Efficacy Endpoint | |
| 8.3.3 | Primary Efficacy Analysis | 26 |
| 8.3.4 | Additional Analyses of the Primary Efficacy Endpoint(s) | 27 |
| 8.4 | Secondary Efficacy Analyses | |
| 8.4.1 | Secondary Efficacy Analyses | |

# Risankizumab M16-011 – Statistical Analysis Plan Version 6.0 – 23 November 2020

| 8.4.2 | Supportive Non-Radiographic Secondary Efficacy Analyses | 30 |
|---|---|---|
| 8.5 | Additional Efficacy Analyses | 31 |
| 8.6 | Efficacy Subgroup Analyses | 34 |
| 9.0 | Safety Analyses | 35 |
| 9.1 | General Considerations | 35 |
| 9.2 | Adverse Events | 37 |
| 9.2.1 | Analysis of Adverse Events for Period 1 | 37 |
| 9.2.1.1 | Adverse Event Overview | 37 |
| 9.2.1.2 | Adverse Events by System Organ Class and Preferred Term | 38 |
| 9.2.1.3 | Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation | 39 |
| 9.2.1.4 | Frequent (≥ 1%) Adverse Events by Preferred Term in Decreasing Frequency | 39 |
| 9.2.1.5 | Areas of Safety Interest | 39 |
| 9.2.2 | Analysis of Adverse Events for Long-Term | 40 |
| 9.2.2.1 | Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure | 40 |
| 9.2.2.2 | Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT | 40 |
| 9.2.2.3 | Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation | 41 |
| 9.2.2.4 | Areas of Safety Interest Rates per 100 Patient-Years of Study Drug Exposure | 41 |
| 9.3 | Analysis of Laboratory Data | 41 |
| 9.3.1 | Variables and Units | 42 |
| 9.3.2 | Analysis of Laboratory Data for Period 1 | 43 |
| 9.3.2.1 | Assessment of Mean Change from Baseline in Clinical Laboratory Variables | 44 |
| 9.3.2.2 | Assessment of Shift from Baseline in Clinical Laboratory Variables | 44 |
| 9.3.2.3 | Assessment of Potentially Clinically Significant Laboratory Values | 45 |
| 9.3.2.4 | Assessment of Liver Function Test Elevations | 45 |
| 9.3.3 | Analysis of Long-Term Laboratory Data | 47 |

# Risankizumab M16-011 – Statistical Analysis Plan Version 6.0 – 23 November 2020

| 9.3.3.1 | Assessment of Mean Change from Baseline in Clinical Laboratory Variables | 47 |
|---|---|---|
| 9.3.3.2 | Assessment of Potentially Clinically Significant Laboratory | |
| | Values | 48 |
| 9.3.3.3 | Assessment of Liver Elevations | 48 |
| 9.4 | Analysis of Vital Signs | 48 |
| 9.4.1 | Analysis of Vital Sign for Period 1 | 49 |
| 9.4.2 | Analysis of Long-Term Vital Sign | 49 |
| 10.0 | Other Analyses | 49 |
| 11.0 | Interim Analyses | 49 |
| 11.1 | Data Monitoring Committee | 49 |
| 12.0 | Overall Type-I Error Control | 50 |
| 13.0 | Version History | |
| 14.0 | References | |
| List of Tab | oles | |
| Table 1. | Subgroups for Efficacy Analysis | 34 |
| Table 2. | List of Laboratory Variables | 42 |
| Table 3. | SAP Version History Summary | 52 |
| List of Fig | ures | |
| Figure 1. | Study Schematic | 8 |
| Figure 2. | An Example of eDISH Plot | 47 |
| Figure 3. | Graphical Testing Procedure | 51 |
| List of App | pendices | |
| Appendix A. | Protocol Deviations | 56 |
| Appendix B. | Definition of Areas of Safety Interest | 57 |
| Appendix C. | Potentially Clinically Significant Criteria for Safety Endpoints | 58 |
| Appendix D. | Definition of Estimand for Primary and Ranked Secondary | |
| | Endpoints | 60 |



Risankizumab
M16-011 – Statistical Analysis Plan
Version 6.0 – 23 November 2020

| Appendix E. | NRI-C Procedure | 62 |
|---|---|---|
| Appendix F. | Tipping Point Analysis for Non-Radiographic Endpoints | 66 |
| Appendix G. | Details of Supplementary Analyses for Radiographic Continuous | |
| | Endpoints | 69 |
| Appendix H. | CTCAE Grades | 73 |
| Appendix I. | Geographic Region | 74 |
| 11 | | |



#### 1.0 Introduction

This Statistical Analysis Plan (SAP) describes the statistical analyses for risankizumab Study M16-011 "A Phase 3, Randomized, Double-Blind Study Comparing Risankizumab to Placebo in Subjects with Active Psoriatic Arthritis (PsA) Who Have a History of Inadequate Response to or Intolerance to at Least One Disease Modifying Anti-Rheumatic Drug (DMARD) Therapy." It provides details to further elaborate statistical methods as outlined in the protocol and describes analysis conventions to guide the statistical programming work.

The analyses of pharmacokinetics/pharmacodynamics, pharmacogenetic, and selected biomarkers will not be covered in this SAP.

Unless noted otherwise, all analyses will be performed using SAS Version 9.4 (SAS Institute Inc., Cary, NC 27513) or later under the UNIX operating system.

# 2.0 Study Design and Objectives

# 2.1 Objectives

# **Primary Objective**

#### **Period 1 Double-Blind**

To compare the efficacy of risankizumab 150 mg versus placebo for the treatment of signs and symptoms of PsA in the study population.

#### **Secondary Objectives**

#### **Period 1 Double-Blind**

1. To compare the efficacy of risankizumab 150 mg versus placebo for the inhibition of progression of structural damage as assessed by radiographs in the study population.



2. To compare the safety and tolerability of risankizumab 150 mg versus placebo in the study population.

#### Period 2 Open-Label

To evaluate the long-term safety, tolerability and efficacy of risankizumab 150 mg in subjects with PsA who have completed Period 1.

# 2.2 Study Design Overview

This is a Phase 3, global, multicenter study that will evaluate subjects with moderate to severely active PsA who have had an inadequate response or intolerance to 1 or more DMARDs (DMARD-IR).

The study consists of a Screening Period (approximately 35 days), Period 1, Period 2, and a 20-week Follow-up Period. Period 1 is a 24-week randomized, double-blind, placebo-controlled, parallel-group period. At Week 24, Period 2 begins. To maintain the blind to original allocation, treatment at the Week 24 Visit will be blinded: subjects randomized to placebo will receive blinded risankizumab 150 mg, and subjects randomized to risankizumab will receive blinded placebo. At Week 28 and for the remaining dosing visits (up to Week 208), all subjects will receive open-label risankizumab 150 mg every 12 weeks. Subjects will remain blinded to the original randomization allocation for the duration of study.

A schematic of the study is shown in Figure 1.

Figure 1. Study Schematic



#### LEGEND:

BL = Baseline; RCT = randomized controlled trial; W = Week

- \* At Week 24, subjects randomized to placebo in Period 1 will receive a blinded dose of risankizumab. Subjects randomized to risankizumab treatment in Period 1 will receive a blinded dose of placebo.
- \*\* At Week 28, subjects randomized to placebo in Period 1 will receive a 2<sup>nd</sup> dose of risankizumab. Subjects randomized to risankizumab in Period 1 will receive risankizumab (scheduled dose).
- \*\*\* From Week 40 and up to Week 208 Visits, doses occur q12w.
- † Follow-up phone call.
  - Dosing
- → Bilateral radiographs. Depending on response at Week 12 and Week 16, radiographs at Week 16 will not apply to all subjects.
- a. At Week 16, subjects classified as non-responders (defined as not achieving at least a 20% improvement in either or both tender joint count [TJC] and swollen joint count [SJC] at both Week 12 and Week 16 compared to Baseline) will have the option to add or modify rescue concomitant medications/therapy as described in Section 5.4 of the study protocol. Rescue therapy qualification occurs only at Week 16 Visit.
- b. Starting at Week 36, subjects classified as non-responders will be discontinued from study drug. See Section 5.5 of the study protocol for details.

The Primary Analysis will be conducted after all ongoing subjects have completed Week 24 and an interim database lock (Week-24 Database Lock) has occurred, to support an interim CSR for the initial regulatory submission. An additional interim database lock will be conducted to provide further efficacy and safety exposure for integrated



summaries of efficacy and safety supporting the initial regulatory submission; no interim CSR will be generated based on this interim lock. After then, additional interim analyses may be conducted as deemed appropriate. The final analysis will be performed after all ongoing subjects complete the study.

#### 2.3 Treatment Assignment and Blinding

Subjects will be randomized to risankizumab 150 mg or placebo in a 1:1 ratio. Randomization will be stratified by extent of psoriasis ( $\geq$  3% BSA or < 3% BSA), current use of at least 1 conventional synthetic disease modifying anti-rheumatic drugs (csDMARD) (0 vs  $\geq$  1), presence of dactylitis (yes vs no), and presence of enthesitis (yes vs no).

### 2.4 Sample Size Determination

Approximately 880 subjects will be randomized to risankizumab 150 mg or placebo in a ratio of 1:1 (440 subjects/treatment group). This sample size provides at least 90% power to detect at least 25% difference in ACR20 response rate (assuming a placebo ACR20 response rate of 35.7%). With the given sample size, there is approximately 80% power to detect a standardized effect size of 0.20 in change from Baseline in PsA-mTSS for risankizumab versus placebo group at Week 24. All power and sample size were calculated based on at two-sided significance level of 0.05 and accounting for a 10% dropout rate.

# 3.0 Endpoints

# 3.1 Primary Endpoint(s)

The primary endpoint is ACR20 response at Week 24.

# 3.2 Secondary Endpoint(s)

The following is a list of ranked secondary endpoints with multiplicity adjustment:



- Change from Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) score at Week 24;
- Psoriasis Area Severity Index (PASI) 90 response at Week 24 (for subjects with BSA ≥ 3% at Baseline);
- 3. ACR20 response at Week 16;
- 4. Minimal Disease Activity (MDA) response at Week 24;
- 5. Change from Baseline in modified Nail Psoriasis Severity Index (mNAPSI) scores at Week 24 (for subjects with nail psoriasis at baseline);
- 6. Change from Baseline in in Physician's Global Assessment of Fingernail Psoriasis (PGA-F) (for subjects with nail psoriasis at baseline);
- 7. Resolution of enthesitis defined as Leeds Enthesitis Index (LEI) = 0 at Week 24 (for subjects with baseline presence of enthesitis (LEI > 0) pooled from M15-998 and M16-011);
- 8. Resolution of dactylitis defined as Leeds Dactylitis Index (LDI) = 0 at Week 24 (for subjects with baseline presence of dactylitis (LDI > 0) pooled from M15-998 and M16-011);
- 9. Change from Baseline in modified Total Sharp Score (PsA-mTSS) at Week 24;
- 10. Change from Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) scores at Week 24;
- 11. Change from Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) scores at Week 24.

Other secondary endpoints without multiplicity adjustment are:

- 1. ACR50 response at Week 24;
- 2. ACR70 response at Week 24.



#### 3.3 Additional Efficacy Endpoints

Additional efficacy endpoints at all scheduled visits (when measurements are collected) are listed below.

- ACR20/50/70 response;
- No radiographic progression response (defined as change from Baseline in PsA-mTSS ≤ 0) at Week 24, Week 52, and Week 100;
- No radiographic progression response (defined as change from Baseline in PsA-mTSS ≤ 0.5) at Week 24, Week 52, and Week 100;
- Change from Baseline in joint space narrowing score (JSN) and joint erosion score (JES), as assessed by radiographs at Week 24, Week 52, and Week 100;
- Change from Baseline in individual components of ACR response;
  - $\circ$  Change from Baseline in Tender Joint Count (TJC) (0-68);
  - $\circ$  Change from Baseline in Swollen Joint Count (SJC) (0-66);
  - Change from Baseline in Physician Global Assessment of Disease Activity
     (PGA) (mm on a 100-mm horizontal visual analogue scale [VAS]);
  - Change from Baseline in Patient's Global Assessment of Disease Activity (PtGA) (mm on a 100-mm horizontal visual analogue scale [VAS]);
  - Change from Baseline in Patient's Assessment of Pain (mm on a 100-mm horizontal visual analogue scale [VAS]);
  - Change from Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) score;
  - Change from Baseline in High-Sensitivity C Reactive Protein (hs-CRP);
- MDA response;
- Change from Baseline in LDI (for subjects with baseline LDI > 0);
- Change from Baseline in dactylitis count (for subjects with baseline LDI > 0)
- Resolution of dactylitis (LDI = 0) (for subjects with baseline LDI > 0);
- Change from Baseline in LEI (for subjects with baseline LEI > 0);
- Resolution of enthesitis (LEI = 0) (for subjects with Baseline LEI > 0);



- Change from Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index (for subjects with baseline SPARCC Enthesitis Index > 0);
- Resolution of enthesitis sites included in the SPARCC Enthesitis Index (for subjects with baseline SPARCC Enthesitis Index > 0);
- Change from Baseline in total enthesitis count (for subjects with baseline LEI > 0 and baseline SPARCC Enthesitis Index > 0);
- Resolution of enthesitis in both LEI and SPARCC (defined as LEI = 0 and SPARCC = 0) (for subjects with baseline LEI > 0 and baseline SPARCC Enthesitis Index > 0)
- PASI 75/90/100 response (for subjects with BSA  $\geq$  3% at baseline);
- Achievement of both PASI90 and ACR50 (for subjects with BSA ≥ 3% at baseline);
- Change from Baseline in BSA-PsO in subjects with BSA  $\geq$  3% at baseline;
- Modified Psoriatic Arthritis Response Criteria (PsARC) response;
- Change from Baseline in Disease Activity Score 28 using high sensitivity C-Reactive Protein (DAS28-hsCRP);
- Change from Baseline in PsA Disease Activity Score (PASDAS);
- Change from Baseline in Disease Activity in Psoriatic Arthritis (DAPSA) score;
- Change from Baseline in the FACIT-Fatigue Questionnaire score;
- Change from Baseline in SF-36 Health Questionnaire physical component summary, mental component summary and the 8 sub-domain scores;
- Change from Baseline in EuroQol-5D-5L (EQ-5D-5L) Health Questionnaire index and VAS score;
- Change from Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire measures;
- Health resource utilization (HRU) since the last study visit;
- Change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score (for subjects with spondylitis at baseline, for subjects with spondylitis at Baseline confirmed by radiography or MRI);



- Change from Baseline in modified BASDAI score (for subjects with spondylitis at Baseline, for subjects with spondylitis at Baseline confirmed by radiography or MRI);
- Change from Baseline in BASDAI Spinal Pain (for subjects with spondylitis at Baseline, for subjects with spondylitis at Baseline confirmed by radiography or MRI);
- BASDAI 50 response (for subjects with spondylitis at Baseline and for subjects with spondylitis at Baseline confirmed by radiography or MRI);
- Change from Baseline in morning stiffness score (mean of BASDAI Questions 5 and 6) (for subjects with spondylitis at Baseline, for subjects with spondylitis at Baseline confirmed by radiography or MRI);
- Change from Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) (for subjects with spondylitis at baseline and for subjects with spondylitis at Baseline confirmed by radiography or MRI);
- ASDAS Inactive Disease (for subjects with spondylitis at baseline and for subjects with spondylitis at Baseline confirmed by radiography or MRI);
- ASDAS Major Improvement (for subjects with spondylitis at baseline and for subjects with spondylitis at Baseline confirmed by radiography or MRI);
- ASDAS Clinically Important Improvement (for subjects with spondylitis at baseline and for subjects with spondylitis at Baseline confirmed by radiography or MRI);
- Change from Baseline in PGA-F score (for subjects with nail psoriasis at baseline);
- Achievement of PGA-F score of 'clear' or 'minimal' with at least a 2-grade improvement (for subjects with 'mild' 'moderate' or 'severe' at baseline)
- Change from Baseline in mNAPSI score (for subjects with nail psoriasis at baseline);
- Achievement of a clinically meaningful improvement in HAQ-DI scores defined as  $\Delta$ HAQ-DI  $\leq$  -0.35 (for subjects with HAQ-DI  $\geq$  0.35 at baseline).



#### 3.4 Safety Endpoints

Safety evaluations include adverse event (AE) monitoring, physical examinations, vital sign measurements, and clinical laboratory testing (hematology and chemistry) as a measure of safety and tolerability for the entire study duration.

#### 3.5 Additional Endpoints

No additional endpoints will be analyzed in the SAP. Pharmacological parameters will be analyzed separately and is not included in this SAP.

# 4.0 Analysis Populations

The Full Analysis Set (FAS) includes all randomized subjects who received at least one dose of study drug. The FAS will be used for all efficacy and baseline analyses. Subjects will be included in the analysis according to the treatment groups that they are randomized to.

The Per-Protocol Analysis Set consists of a subset of FAS subjects who did not have any major protocol deviations that are determined to have a potential impact on the primary efficacy endpoint up to Week 24 in Period 1 of the study. Additional analysis of the primary efficacy endpoint will be conducted on the Per-Protocol Analysis Set.

The final criteria and the exclusion of subjects for the Per-Protocol Analysis will be identified prior to Primary Analysis database lock.

The Safety Analysis Set consists of all subjects who received at least one dose of study drug. Subjects will be included in the analysis according to the study drug that they actually received. The Safety Analysis Set will be used for all safety analysis.

# 5.0 Subject Disposition

The total number of subjects who were randomized and who were treated will be summarized.



A summary of subject accountability will be provided where the number of subjects in each of the following categories will be summarized for each randomized treatment group:

- Subjects randomized in the study;
- Subjects included in key analysis populations (FAS, Per Protocol Analysis Set, Safety Analysis Set);
- Subjects who took at least one dose of study drug;
- Subjects who completed Period 1 study participation;
- Subjects who entered Period 2;
- Subjects who completed overall study (Period 1 and Period 2) participation;
- Subjects who prematurely discontinued study drug (all reasons and primary reason);

For end of study participation, the number and percentage of subjects who completed the protocol defined follow-up period (or did not with associated reasons) will be summarized overall and by treatment group.

# 6.0 Study Drug Duration and Compliance

For the Safety Analysis Set, duration of treatment will be summarized for risankizumab 150 mg and placebo for Period 1, and for risankizumab 150 mg for long-term. Duration of treatment is defined for each subject as last dose date - first dose date + 84 days. Duration of treatment will be summarized using the number of subjects treated, mean, standard deviation, median, minimum and maximum.

Treatment compliance will be summarized by treatment group at Week 24 for the FAS population. Treatment compliance is defined as the number of injections administered during the subject's participation up to Week 24 divided by the number of injections planned during the subject's participation in the treatment phase up to Week 24. Compliance will be calculated for each subject and summarized with the mean, median, standard deviation, minimum, and maximum.



# 7.0 Demographics, Baseline Characteristics, Medical History, and Prior/Concomitant Medications

Demographics, baseline or disease characteristics, medical history, and prior and concomitant medications will be summarized for the FAS by treatment group and overall. Categorical variables will be summarized with the number and percentage of subjects. Continuous variables will be summarized with descriptive statistics (number of non-missing observations, mean and standard deviation, median, minimum and maximum).

# 7.1 Demographics and Baseline Characteristics

The following demographic and baseline characteristics will be summarized.

#### **Demographic Characteristics**

- Sex (male, female)
- Age (years)
- Age Categories ( $<65, \ge 65 \text{ years}, \ge 65 \text{ years}$  and  $<75, \ge 75 \text{ years}$ )
- Race (White, Black or African American, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Asian, Other)
- Geographic Region (North America, South/Central America, Western Europe, Eastern Europe, Asia, Other)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
- Weight (kg)
- Weight Categories ( $< 100 \text{ kg}, \ge 100 \text{ kg}$ )
- Height (cm)
- Body Mass Index (BMI) (kg/m<sup>2</sup>)
- Body Mass Index (BMI) Category (kg/m<sup>2</sup>) ( $< 25, \ge 25$  and  $< 30, \ge 30$ )

#### **PsA Medical History and Prior and Concomitant Medications**

• Duration of PsA in years



- Duration of PsA in years Categories ( $\leq 5$ ,  $\geq 5$  and  $\leq 10$ ,  $\geq 10$  years)
- Number of prior csDMARDs  $(0, 1, 2, \ge 3)$
- Nonsteroidal anti-inflammatory drug (NSAID) use at baseline (yes, no)
- Oral Corticosteroid use at baseline (yes, no)
- Concomitant MTX use at baseline (yes, no)
- Concomitant csDMARD at baseline

#### Any csDMARD

- o Any MTX
  - MTX alone
  - MTX and other csDMARD
- o csDMARD other than MTX
  - Any sulfasalazine, without MTX
  - Any leflunomide, without MTX
  - Any apremilast, without MTX

None

#### **Baseline Disease Characteristics**

#### Categorical:

- MDA (Minimal Disease Activity) for PsA (yes, no)
- Presence of Dactylitis based on LDI (LDI > 0) (yes, no)
- Presence of Enthesitis based on LEI (LEI > 0) (yes, no)
- Presence of Enthesitis based on SPARCC (SPARCC Enthesitis Index > 0) (yes, no)
- Presence of nail psoriasis (yes, no)
- Body Surface Area (BSA) of psoriatic plaques ( $\geq 3\%$ , < 3%)
- Presence of spondylitis (yes, no)
- Anti-cyclic citrullinated peptide (Anti-CCP) status (Positive (≥ 17 U/mL), Negative (< 17 U/mL))</li>



- Rheumatoid Factor (RF) status (Positive (≥ 15 IU/mL), Negative (< 15 IU/mL))</li>
- Categories for hsCRP ( $< 3.0, \ge 3.0 \text{ mg/L}$ )

#### Continuous

- PASI Psoriasis Area and Severity Index (PASI) (for subjects with BSA ≥ 3% at Baseline)
- Modified Total Sharp Score (PsA-mTSS)
- Disease Activity Score in 28 joints hsCRP (DAS28 (CRP))
- Total dactylitis count (for subjects with presence of dactylitis (LDI > 0))
- LDI (for subjects with presence of dactylitis (LDI > 0))
- Total enthesitis count (for subjects with presence of enthesitis (total enthesitis count > 0))
- LEI (for subjects with LEI > 0)
- Classification Criteria for PsA (CASPAR classification criteria total score)
- BSA of psoriatic plaques (BSA-PsO) (for subjects with BSA  $\geq$  3% at Baseline and for all subjects)
- SPARCC Enthesitis Index (for subjects with SPARCC Enthesitis Index > 0)
- Modified Nail Psoriasis Severity Index (mNAPSI) score (for subjects with nail psoriasis at baseline; score range: 0 – 130)
- Physician's Global Assessment of Fingernail Psoriasis score (PGA-F) (for subjects with nail psoriasis at baseline; score range: 0-4)
- Tender joint count (TJC68) defined as the number of tender joints out of 68 assessed joints
- Swollen joint count (SJC66) defined as the number of swollen joints out of 66 assessed joints
- Tender joint count (TJC28) defined as the number of tender joints out of 28 assessed joints used for DAS28 calculation
- Swollen joint count (SJC28) defined as the number of swollen joints out of 28 assessed joints used for DAS28 calculation



- Physician's global assessment of disease activity (mm on a 100-mm horizontal visual analogue scale [VAS])
- Patient's assessment of pain score (mm on a 100-mm horizontal VAS)
- Patient's global assessment of disease activity score (mm on a 100-mm horizontal VAS)
- Health Assessment Questionnaire Disability Index (HAQ DI) scores
- High sensitivity C-reactive protein (hsCRP) (mg/L)
- Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) score
- 36-Item Short Form Health Survey (SF-36) Version 2: physical component summary, mental component summary and the 8 sub-domain scores
- EurQol-5d-5L (EQ-5D-5L) index and VAS score
- Work Productivity and Activity Impairment (WPAI) measures
- Bath Ankylosing Spondylitis Activity Index (BASDAI) score (for subjects with spondylitis at Baseline, for subjects with spondylitis at Baseline confirmed by radiography or MRI)
- Modified BASDAI score (for subjects with spondylitis at Baseline, for subjects with spondylitis at Baseline confirmed by radiography or MRI)
- BASDAI Spinal Pain (for subjects with spondylitis at Baseline, for subjects with spondylitis at Baseline confirmed by radiography or MRI)
- ASDAS score (for subjects with spondylitis at Baseline, for subjects with spondylitis at Baseline confirmed by radiography or MRI)

#### **Tobacco/Nicotine and Alcohol Use**

- Tobacco/Nicotine Use (current, former, never, unknown)
- Alcohol Use (current, former, never, unknown)

# 7.2 Medical History

Medical history data will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The actual version of the MedDRA coding dictionary will be noted in the



statistical tables and clinical study report. The number and percentage of subjects in each medical history category (by MedDRA system organ class and preferred term) will be summarized overall and by treatment group. The system organ class (SOC) will be presented in alphabetical order, and the preferred terms will be presented in alphabetical order within each SOC. Subjects reporting more than one condition/diagnosis will be counted only once in each row (SOC or preferred term).

#### 7.3 Prior and Concomitant Medications

Prior and concomitant medications will be summarized by generic name. A prior medication is defined as any medication taken prior to the date of the first dose of study drug (risankizumab or placebo). A concomitant medication is defined as any medication that started prior to the date of the first dose of study drug and continued to be taken after the first dose of study drug or any medication that started on or after the date of the first dose of study drug, but not after the date of the last dose of study drug + 140 days. The number and percentage of subjects taking medications will be summarized by generic drug name based on the World Health Organization (WHO) Drug Dictionary for both prior and concomitant medications. In addition, the number and percentage of subjects taking rescue medication will be summarized by ATC classification level 2, generic drug name and route of administration. A listing of subjects taking rescue medication with generic drug name, dosage and route of administration will also be provided.

# 8.0 Efficacy Analyses

#### 8.1 General Considerations

All efficacy analyses will be conducted in the FAS Population in each period. In addition, Per-protocol analysis for primary endpoint will be performed. All tests will be 2-sided at an alpha level of 0.05.

The Primary Analysis will be conducted after all ongoing subjects have completed Week 24 and the Week-24 Database Lock has occurred. Efficacy and safety analyses will be performed for Period 1 and long-term efficacy and safety will be summarized through



the data cutoff date. An additional interim database lock will be conducted to provide further efficacy and safety exposure for integrated summaries of efficacy and safety supporting the initial regulatory submission; no study-specific analysis will be performed based on this database lock.

Unless otherwise specified, categorical variables will be analyzed using Cochran-Mantel-Haenszel (CMH) test, adjusting for the stratification factors. Continuous variables will be analyzed using Mixed-Effect Model Repeat Measurement (MMRM) method.

Unless otherwise specified, any subject who is randomized based on a wrong stratum will be analyzed according to the actual stratum the subject belongs to.

"Baseline" refers to the last non-missing observation before the first administration of study drug or randomization if no study drug is given.

#### Efficacy analysis for Period 1

The efficacy analysis for Period 1 will be performed after all ongoing subjects have completed Period 1 and an interim database lock has occurred. This is the only and final efficacy analysis in Period 1.

#### Long-term efficacy analysis

Long-term efficacy will be summarized based on data in Period 1 and Period 2 up to data cutoff date for the Week-24 Database Lock. After the initial regulatory submission, additional interim analyses will be performed as deemed appropriate, for example, to address requests from regulatory agencies. The final analysis will be performed after all ongoing subjects complete the study.

Long-term efficacy analysis will be performed on As Observed data (defined in Section 8.2) by randomized treatment group sequence as described below:

1. Placebo → risankizumab 150 mg



#### 2. risankizumab 150 mg → risankizumab 150 mg

There will be no statistical testing for long-term non- radiographic efficacy analysis; only descriptive statistics and 95% confidence intervals will be provided. Nominal p-value will be provided for long-term radiographic efficacy analysis.

#### 8.2 Handling of Missing Data and Intercurrent Events

Missing data could occur due to various reasons, including missing visits/assessments, early withdrawal from the study, or missing due to COVID-19 infection or logistic restriction.

The COVID-19 pandemic is interfering with the conduct of many ongoing trials, with potential impacts on treatment duration and the collection, analysis and the interpretation of clinical trial data. Some protocol-specified visits in the clinical trials may be impacted due to COVID-19 infection or logistical restrictions during the pandemic. For example, some scheduled visits may be missed due to self-quarantine or local government restrictions on travel; some visits may also be delayed or canceled due to healthcare resource constraints during the pandemic. Impacted visits due to COVID-19 will be recorded in the database. The probability of having missed visits and missing data due to COVID-19 infection or logistical restrictions related to the COVID-19 pandemic can be reasonably assumed to be unrelated to the unobserved values. Therefore, for the purpose of statistical analysis, it is reasonable to assume that these missing data are missing at random (MAR) and the statistical models that require MAR assumption are appropriate. The intent is to provide reliable estimates of the treatment effects targeted in the protocol under the scenario without the impact of COVID-19 pandemic. Sensitivity analyses will be performed to assess the impact of missing data and the robustness of the conclusion. Number of subjects with missing values due to COVID-19 will be presented.

Intercurrent events include initiation of rescue medications or initiation of concomitant medications for PsA that could meaningfully impact efficacy assessment. Missing data



and intercurrent events will be handled using the following methods for the efficacy analysis.

# Non-Responder Imputation (NRI) incorporating Multiple Imputation (MI) to handle missing data due to COVID-19 (NRI-C)

The NRI-C data handling will be used for the primary estimand (refer to Section 8.3.1) for the binary variables. This approach will handle missing data for binary variables as follows.

- a. Missing data due to COVID-19 infection or logistical restriction related to COVID-19 pandemic will be handled by MI.
- b. Subject who does not have evaluation during a specific visit window due to reasons other than COVID-19 infection or logistical restriction related to COVID-19 pandemic will be handled by NRI for that visit. NRI will consider a subject with missing evaluation as a non-responder with the exception for composite binary endpoints including ACR20, ACR50, ACR70, MDA and modified PsARC for which the missing components will be imputed with last observation carry forward to derive composite score before imputing missing evaluations as a nonresponder.

Subjects will be considered as non-responders after initiation of rescue medications or initiation of concomitant medications for PsA that could meaningfully impact efficacy assessment; these medications will be identified prior to database lock and unblinding.

For composite binary endpoints including ACR20, ACR50, ACR70, MDA and modified PsARC, the missing binary values due to COVID-19 infection or logistical restriction will be imputed via MI with the logistic regression option as outlined in Appendix F. For other binary endpoints which are dichotomized from a continuous scale, the MI will be applied to the original continuous scale and the dichotomized variable will be derived from the imputed value for missing due to COVID-19 infection or logistical restriction.



#### **Mixed-Effect Model Repeated Measurements (MMRM)**

The repeated measures analysis will be conducted using a mixed model including observed measurements at all visits. For the MMRM analysis, data collected after initiation of concomitant medications for PsA that could meaningfully impact efficacy assessment or initiation of rescue therapy will be excluded. The mixed model includes the categorical fixed effects of treatment, visit and treatment-by-visit interaction, stratification factors, and the continuous fixed covariate of baseline measurement. An unstructured variance covariance matrix will be used. Parameter estimation is based on the assumption of data being missing at random and using the method of restricted maximum likelihood (REML). The MMRM approach is appropriate in handling missing data due to COVID-19 infection or logistical restriction given the validity of the missing at random assumption. MMRM will be used for the primary estimand of continuous variables (refer to Section 8.4.1).

#### As Observed (AO)

The AO analysis will not impute values for missing evaluations, and thus a subject who does not have an evaluation on a scheduled visit will be excluded from the AO analysis for that visit. Regardless of premature discontinuation of study drug, initiation of concomitant medications for PsA that could meaningfully impact efficacy assessment or initiation of rescue medications, all observed data will be used in the analysis. The AO analysis will be used to facilitate the supplementary analysis.

#### **AO** with Imputation

The AO with imputation will use all observed data regardless of premature discontinuation of study drug, initiation of concomitant medications for PsA that could meaningfully impact efficacy assessment or initiation of rescue medications and will impute missing as non-responders. It will be used for the supplementary analysis for binary variables.



#### **Multiple Imputation (MI)**

As a sensitivity analysis, MI will be utilized for both hypothetical and treatment policy estimand (Appendix D). The MI analysis will impute missing data multiple times under appropriate random variation and thus generate multiple imputed "pseudo-complete" datasets. SAS PROC MI will be used to generate 30 datasets using the fully conditional specification (FCS) method. Specifically, treatment group is included in the FCS imputation model to enable stratified sampling. Additionally, the imputation model includes demographics variables and baseline disease characteristics, stratification factors, as well as longitudinal response observed at all other visits. Analysis using CMH for binary endpoints and analysis of covariance (ANCOVA) for continuous endpoints will be performed on each of the multiple imputed datasets. Subsequently SAS PROC MIANALYZE will be used to aggregate the results for the final statistical inference using Rubin's method<sup>5</sup>.

#### **Linear Extrapolation for Radiographic Data**

For radiographic data (e.g., mTSS-based endpoints), linear extrapolation will be applied to subjects with missing data or subjects who prematurely discontinued study drug or received rescue medication, where the radiographic data at the time point of interest (e.g., Week 24/52) will be imputed with data from prior visits assuming a linear relationship. Linear extrapolation will be used to facilitate the primary estimand for radiographic endpoints (refer to Section 8.4.1).

#### 8.3 Primary Efficacy Endpoint and Analysis

#### 8.3.1 Primary Efficacy Endpoint

The primary efficacy endpoint is ACR20 response at Week 24. The attributes of primary estimand based on composite estimand framework are outlined in Appendix D.



# 8.3.2 Handling of Missing Data and Intercurrent Event for the Primary Efficacy Endpoint

For the primary estimand, NRI-C as defined in Section 8.2 will be used.

Subjects who initiated concomitant medications for PsA that could meaningfully impact efficacy assessment or were rescued prior to Week 24 or missed ACR20 response at Week 24 will be treated as non-responders. The number and percentage of non-responders for ACR20 will be summarized into one of the five categories for which the episode occurs first:

- 1. Subjects who were rescued before Week 24
- 2. Subjects who initiated concomitant medications for PsA that could meaningfully impact efficacy assessment by Week 24
- 3. Subjects with ACR20 measurements observed at Week 24 but did not meet ACR20 response criteria
- 4. Subjects with missing Week 24 ACR20 measurements due to the reasons other than COVID-19 infection or logistical restriction related to COVID-19 pandemic
- 5. Subjects with missing Week 24 ACR20 measurements due to COVID-19 infection or logistical restriction related to COVID-19 pandemic

# 8.3.3 Primary Efficacy Analysis

Analysis of the primary endpoint will be conducted on the FAS based on randomized treatment group (risankizumab 150 mg versus placebo) using NRI-C for missing data handling. Point estimate and 95% CI using normal approximation will be provided for the response rate for each randomized treatment group. Comparisons of the primary endpoint will be made between the risankizumab and placebo group using the CMH adjusting for stratification factors. Point estimate, 95% CI and nominal p-value for the treatment comparison will be presented. Refer to Appendix E for the details of NRI-C procedure and respective statistical inference.



A sensitivity analysis will be conducted on the Per Protocol Analysis Set using the CMH model and NRI-C missing data handling.

#### 8.3.4 Additional Analyses of the Primary Efficacy Endpoint(s)

For the primary efficacy endpoint, a supplementary analysis will be based on treatment policy estimand framework using the same CMH method and AO data. The attributes of the corresponding estimand are outlined in Appendix D.

For the treatment policy estimand, additional supplementary analysis will be conducted using AO with imputation. The same CMH method will be conducted.

Additional supplementary analyses using MI as outlined in Section 8.2 based on AO data, i.e., all observed data regardless of study drug adherence, concomitant medications use for PsA or rescue, will also be conducted to handle missing ACR20 responses. To assess the deviation from missing at random (MAR) assumptions, tipping point analysis will be conducted as a sensitivity analysis for this supplementary analysis. Details of the analysis are outlined in Appendix F.

The assigned treatment information on several subjects was inadvertently shared with the Study project manager (SPM). The blind was restored immediately upon discovery. There was no unblinding to the subjects or investigators nor to the sponsor personnel engaged in the scientific analysis of the study. However, conservatively, a sensitivity analysis for primary endpoint excluding those unblinded subjects from Full Analysis Set will also be performed.

# 8.4 Secondary Efficacy Analyses

# 8.4.1 Secondary Efficacy Analyses

The secondary endpoints are defined in Section 3.2. Ranked secondary endpoints will be tested in rank order, according to procedures in Section 12.0. Resolution of enthesitis and dactylitis will be analyzed as ranked secondary endpoints using pooled data from both M15-998 and M16-011.



For all binary secondary endpoints, frequencies and percentages will be reported for each treatment group. The primary estimand and analysis method are the same as that for the primary efficacy endpoint as defined in Section 8.3.1. NRI-C missing data handling will be used to analyze the primary estimand (refer to Appendix E).

For the secondary endpoints applicable only for a sub-population, the estimand will be constructed similarly but based on the sub-population, as defined in the below table.

| Endpoints | Sub-population |
|---|---|
| Psoriasis Area Severity Index (PASI)<br>90 response at Week 24 | Subjects with BSA $\geq$ 3% at baseline are included in the analysis |
| Change from Baseline in modified Nail<br>Psoriasis Severity Index (mNAPSI) at<br>Week 24 | Subjects with nail psoriasis at baseline are included in the analysis |
| Change from Baseline in Physician's<br>Global Assessment of Fingernail<br>Psoriasis (PGA-F) at Week 24 | Subjects with nail psoriasis at baseline are included in the analysis |
| Resolution of enthesitis (LEI = 0) at Week 24 | Subjects with baseline presence of enthesitis (LEI > 0) are included in the analysis |
| Resolution of dactylitis (LDI = 0) at Week 24 | Subjects with baseline presence of dactylitis (LDI > 0) are included in the analysis |

Comparisons of resolution of enthesitis/dactylitis pooled from M15-998 and M16-011 will be made between the risankizumab and placebo group using the CMH adjusting for common stratification factors (extent of psoriasis and current use of csDMARD) and study.

#### Non-Radiographic Continuous Endpoints

For non-radiographic continuous secondary endpoints, primary analysis will be based on the hypothetical estimand. The attributes of the corresponding estimand are outlined in Appendix D. The comparison is risankizumab 150 mg vs placebo for patients randomized and treated with at least one dose of study drug. Statistical inference will be conducted



using the MMRM model and the associated data handling as described in Section 8.2. The least square (LS) mean and 95% CI for each randomized treatment group and the LS mean for treatment difference, the associated 95% CI and the p-value between risankizumab 150 mg group and the placebo group will be provided.

#### Change from baseline in modified Total Sharp Score (mTSS) at Week 24

For change from baseline in modified Total Sharp Score (mTSS) at Week 24, statistical inference will be conducted using the associated data handling (i.e., linear extrapolation) as described in Section 8.2 and ANCOVA model with treatment and the stratification factors and the corresponding baseline values as the covariates. The attributes of primary estimand based on hypothetical estimand framework are outlined in Appendix D. The comparison will be between risankizumab 150 mg vs placebo for patients randomized and treated with at least one dose of study drug.

To incorporate the uncertainty of a single imputation, the Multiple Imputation (MI) analysis will be conducted as a sensitivity analysis. The proposed MI model for the change from baseline in mTSS will be based on the linearity assumption for the subjects with missing data including those due to premature discontinuation of study drug or use of rescue medication. More specifically, the regression method will be used where missing Week 24 observations will be imputed by regression upon all previous visits, stratified by treatment group. The imputation model will also include baseline demographics and key baseline characteristics as appropriate. ANCOVA will be performed on each of the multiple imputed datasets. The results will be aggregated across the multiple imputed datasets using Rubin's method. The detailed SAS procedure is outlined in Appendix G.

A supplementary analysis will be based on treatment policy estimand framework using AO data, i.e., all observed data regardless of study drug adherence or rescue, handled with the same ANCOVA model. The attributes of the corresponding estimand are outlined in Appendix D. The analysis will be conducted for those who are randomized, received study drug and have the efficacy measurement at Week 24 visit. The LS mean and 95% CI for each randomized treatment group and the LS mean treatment difference, the



associated 95% CI and the p-value between two groups will be provided. Additional supplementary analyses using MI may also be conducted to handle missing mTSS in addition to AO data. To assess the deviation from missing at random (MAR) assumptions, tipping point analysis may be conducted as a sensitivity analysis for this supplementary analysis. Details of the analysis are outlined in Appendix G.

In another sensitivity analysis, a random coefficient model will be applied, in which mTSS measurements are used as the response variable, including measurements at Baseline and post-Baseline. The model is specified with a random intercept and a random slope on time, and includes treatment, stratification factors, and treatment-by-time interaction in the model. The "group" option in PROC MIXED is used to allow for heterogeneity among treatment groups in the covariance structure. The coefficient for treatment-by-time interaction is used to estimate the difference in rate of progression (per 24 weeks) comparing risankizumab 150 mg group and placebo. The rate of progression (per 24 weeks) for each group respectively is also estimated using the coefficients for time and treatment-by-time interaction. In case the random coefficient model does not converge, a simplified model may be explored by removing the random intercept or fitting a fixed-effect linear effect model.

Additionally, in the event that data severely deviates from the normal distribution, non-parametric analyses such as the ranked ANCOVA may be considered for treatment comparison.

# 8.4.2 Supportive Non-Radiographic Secondary Efficacy Analyses

For binary secondary endpoints, the same CMH analyses as the supplementary analyses will be conducted using AO and AO with imputation. The corresponding supplementary estimand is the same as defined in Section 8.3.4 except for the definition of the efficacy measurement (refer to Appendix D).

For non-radiographic continuous secondary endpoints, supplementary analyses on the FAS will be performed based on AO using the treatment policy estimand framework



(refer to Appendix D). The statistical inference will be conducted using ANCOVA model including treatment as the fixed factor and the corresponding baseline value and the stratification factors as the covariates. The LS mean and 95% CI will be reported for each randomized treatment group; the LS mean treatment difference and associated 95% CI and p-value will be reported comparing risankizumab 150 mg group with the placebo group.

For HAQ-DI at Week 24, additional supplementary analyses will be conducted using MI as outlined in Section 8.2 based on AO data under MAR assumption. To assess deviations from MAR, the tipping point analyses will also be conducted using MI as additional sensitivity analyses. Details of the MI and tipping point analysis are outlined in Appendix F.

Due to a technical unblinding incident, a sensitivity analysis for change from baseline in HAQ-DI at Week 24 excluding those unblinded subjects from Full Analysis Set will also be performed.

#### 8.5 Additional Efficacy Analyses

Additional endpoints defined in Section 3.3 will be analyzed at scheduled time points other than those specified for the primary and secondary variables.

#### **Additional Efficacy Analyses for Period 1**

#### Non-radiographic Endpoints

Additional endpoints will be analyzed for each randomized treatment group for all visits using similar statistical methods as for the primary and secondary endpoints.

For binary endpoints, point estimate and 95% CI using normal approximation will be provided for the response rate for each randomized treatment group. Point estimate, 95% CI and p-value will be provided for the treatment comparison between risankizumab 150 mg and the placebo group based on the CMH test adjusting for stratification factors.



Only the nominal p-value will be provided. NRI-C for missing data handling will be used. AO analysis will be used as supplementary analysis.

For continuous endpoints, the LS-mean and 95% CI will be reported for each randomized treatment group. The LS mean treatment difference and associated 95% CI and p-values between risankizumab 150 mg and the placebo group will be provided using MMRM model. Only the nominal p-value will be provided. Data observed after initiation of concomitant medications for PsA that could meaningfully impact efficacy assessment or initiation of rescue will be excluded. Supplementary analysis will be conducted based on ANCOVA model using AO data, with treatment and stratification factors as the fixed factors and the corresponding baseline value as the covariates. Nominal p-values will be provided.

For HRU related endpoints, number and percentage of subjects with non-study health visits will be provided by visit and over the Period 1 up to Week 24. In addition, cumulative number of utilizations per time (e.g., subject-year) up to Week 24 will be provided for each category.

#### Radiographic Endpoints

For no radiographic progression endpoint at Week 24, point estimate and 95% CI using normal approximation of the response rate for each randomized treatment group will be provided. Comparisons will be made between treatment group and placebo group using the CMH test adjusting for stratification factors. Point estimate, 95% CI and nominal p-value for the treatment comparison will be presented. Non-progression will be derived using both linear extrapolation imputation and AO.

For change from baseline in joint space narrowing score and joint erosion score at Week 24, linear extrapolation analysis and AO analysis will be performed similarly as described in Section 8.4.1.



#### Efficacy Analyses for Long Term

Assessments to evaluate long-term efficacy will be analyzed for all efficacy measurements at scheduled visits.

#### Non-radiographic Endpoints

Descriptive statistics will be provided for each randomized treatment sequence as defined in Section 8.1. These include the number of observations, mean, standard deviation, 95% CI, median, minimum, and maximum for continuous endpoints; and frequencies and percentages with 95% CI using normal approximation for binary endpoints. Plot for each randomized treatment group sequence over time will be provided for primary and multiplicity-controlled secondary endpoints and selected additional endpoints. These efficacy analyses will be based on AO data analysis.

A similar analysis for HRU endpoints will be provided at Week 52.

#### Radiographic Endpoints

In the linear extrapolation analysis for Week 52 radiographic endpoints, the missing Week 52 data will be imputed via linear extrapolation using available post-baseline radiographic data in the latest analysis window prior to Week 52. For placebo subjects who switch to risankizumab at Week 24 (if not already rescued at Week 16), their Week 52 radiographic data will be imputed via linear extrapolation using Week 24 radiographic data; for placebo subjects who rescued at Week 16, their Week 52 radiographic data will be imputed via linear extrapolation using Week 16 radiographic data. In the AO analysis, the observed Week 52 measurements will be used regardless of treatment switching. Similar statistical inference approach as Week 24 analysis by original randomized treatment group will be used. Nominal p-values will be provided.



# 8.6 Efficacy Subgroup Analyses

The primary efficacy endpoint will be examined in the subgroups listed in Table 1 below. Treatment difference between risankizumab 150 mg and the placebo group in each category of a subgroup will be presented with point estimate and 95% confidence interval using CMH test adjusting for stratification factors. No p-value will be provided for subgroup analysis. Forest plots presenting the treatment effect of all categories of subgroups will be provided.

Table 1. Subgroups for Efficacy Analysis

| Subgroup Factor | Categories |
|---|---|
| Age | $<65, \ge 65 \text{ years}, \ge 65 \text{ years and} < 75, \ge 75 \text{ years}$ |
| Sex | Male vs Female |
| BMI | $< 25, \ge 25 \text{ and } 30, \ge 30 \text{ kg/m}^2$ |
| Race | White vs Non-white |
| Geographic Region | North America, South/Central America, Western<br>Europe, Eastern Europe, Asia, Other |
| Number of prior csDMARDs | ≤ 1 vs > 1 |
| Presence of enthesitis at Baseline based on LEI | yes vs no |
| Presence of dactylitis at Baseline based on LDI | yes vs no |
| C-Reactive Protein at Baseline | $< 3 \text{ vs} \ge 3 \text{ mg/L}$ |
| Extent of psoriasis at Baseline | $\geq$ 3% BSA vs $<$ 3% BSA |
| Duration of PsA | $\leq 5, > 5 \text{ and } \leq 10, > 10 \text{ years}$ |
| Concomitant csDMARD at baseline | Any csDMARD • Any MTX o MTX alone o MTX and other csDMARD • csDMARD other than MTX None |



# 9.0 Safety Analyses

#### 9.1 General Considerations

Safety analyses will be carried out using the Safety Analysis Set. For the safety analysis, subjects are assigned to a treatment group based on the treatment actually received, regardless of the treatment randomized. A subject's actual treatment will be determined by the first dose of study drug that the subject received.

There are two sets of planned safety analysis: safety analysis for Period 1, and long-term safety analysis.

#### **Safety Analysis for Period 1**

Standard safety analysis by the actual treatment groups of risankizumab 150 mg and placebo will be performed on safety data up to Week 24. No protocol-defined treatment switching will occur prior to this time point.

The standard safety analyses will include reporting of adverse events (AEs), laboratory, and vital signs measurements. Frequency tables of subjects with treatment-emergent adverse events (TEAEs) by system organ class (SOC) and by preferred term (PT) as in the Medical Dictionary for Regulatory Activities (MedDRA) dictionary will be provided by treatment group. All continuous laboratory parameters and vital signs variables at each visit will also be summarized by actual treatment group. Frequency tables of subjects meeting criteria for potentially clinically significant vital sign values and for potentially clinically significant laboratory values will be provided by treatment group.

#### **Long-Term Safety Analysis**

Long-term safety analysis will be performed on all cumulative safety data in Period 1 and Period 2 up to data cutoff date for any interim lock as deemed appropriate and final lock.

Long-term safety analyses that account for protocol-defined treatment switching include reporting of AE rate adjusted by cumulative exposure, descriptive summary in laboratory



parameters and vital sign variables, and rate of potentially clinically significant laboratory and vital signs values.

To adjust for potentially different follow-up time between treatment groups, exposure-adjusted event rate (EAER) will be provided for long term safety analysis. The EAER will be presented for Any Risankizumab group by actual treatment received at the time of AE. The Any Risankizumab group includes subjects who started on Risankizumab 150 mg at randomization and who switched from placebo to Risankizumab 150 mg.

For EAER calculation, the numerator will be the total number of AEs reported for the event (i.e., a subject can contribute more than one event to the numerator) and the denominator will be the total exposure time among subjects under the treatment. The number of AEs reported (numerator), the total number of years of study drug exposure (denominator calculated as total number of days exposed to study drug (i.e., last dose date – first dose date + 140 days) for all treated subjects divided by 365.25), and the exposure-adjusted AE event rate per 100 patient-years calculated as ([numerator (number of AEs)/denominator]) • 100 will be presented for each treatment group.

All continuous laboratory parameters and vital signs variables at each visit will be summarized by actual treatment group sequence defined as follows.

- 1. Placebo → Risankizumab 150 mg
- 2. Risankizumab 150 mg → Risankizumab 150 mg

Frequency tables and listings of subjects meeting criteria for potentially clinically significant vital sign values and for potentially clinically significant laboratory values will be provided for Any Risankizumab group by actual treatment received at the time of event. Missing safety data will not be imputed.


#### 9.2 Adverse Events

A treatment-emergent Adverse Event (TEAE) is defined as an adverse event with an onset date that is after the first dose of study drug, and no more than 140 days of the drug after the last dose of study drug.

Adverse events (AEs) will be summarized and presented using primary MedDRA System Organ Classes (SOCs) and preferred terms (PTs) according to the version of the MedDRA coding dictionary used for the study at the time of database lock. The actual version of the MedDRA coding dictionary used will be noted in the AE tables and in the clinical study report. Specific adverse events will be counted once for each subject for calculating percentages, unless stated otherwise. In addition, if the same adverse event occurs multiple times within a subject, the highest severity and level of relationship to investigational product will be reported.

### 9.2.1 Analysis of Adverse Events for Period 1

#### 9.2.1.1 Adverse Event Overview

An overview of AEs will be presented consisting of the number and percentage of subjects experiencing at least one event for each of the following AE categories:

- Any TEAEs
- Any COVID-19 related TEAEs
- Any TEAE related to study drug according to the investigator
- Any serious TEAE
- Any severe TEAE
- Any TEAE leading to discontinuation of study drug
- Any TEAE leading to death
- All deaths
  - o COVID-19 related deaths
  - o Deaths occurring  $\leq 140$  days after last dose of study drug
  - o Deaths occurring > 140 days after last dose of study drug.



Additional AEs may be considered for tabulation/summary based on recommendations from Clinical and Safety as deemed appropriate.

The number and percentage of subjects experiencing at least one event of treatment-emergent AEs will be summarized for each treatment group. The point estimate and 95% CI (using normal approximation and separate group variance) will be provided for the treatment difference in AE percentage between risankizumab group and the placebo group. An overview of the AE of safety interest (ASI) will be provided similarly and the categories of ASI is defined in Section 9.2.1.4. In addition, an overview of AEs per 100 patient-years of study exposure will be presented for the AE categories defined above. The number of TEAEs reported, the total number of years of study drug exposure, and the TEAE rate per 100 patient-years will be presented.

COVID-19 cases will be identified using relevant terms for COVID-19 search available in MedDRA version 23.0 or higher. All COVID-19 related AEs and COVID-19 related deaths will be summarized in the TEAE Overview table.

### 9.2.1.2 Adverse Events by System Organ Class and Preferred Term

Treatment-emergent adverse events will be summarized by SOC and PT, the following summaries of adverse events will be generated:

- All TEAEs
- Serious TEAEs
- Severe TEAEs
- TEAEs related to study drug according to the investigator
- TEAEs leading to discontinuation of study drug
- TEAE leading to death
- COVID-19 related TEAE

Subjects reporting more than one adverse event for a given MedDRA preferred term will be counted only once for that term (most severe incident for the severity tables and most



related incident for the relationship tables). Subjects reporting more than one type of adverse event within a SOC will be counted only once for that SOC. Subjects reporting more than one type of adverse event will be counted only once in the overall total.

TEAEs will also be summarized by relationship to risankizumab 150 mg and placebo, as assessed by the investigator as well as by maximum severity, by treatment groups.

The SOCs will be presented in alphabetical order, and the PTs will be presented in alphabetical order within each SOC.

## 9.2.1.3 Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation

All serious adverse events (SAEs) including deaths and adverse events leading to discontinuation of study drug will be listed in tables, besides summary by SOC and PT covered in Section 9.2.1.2.

# 9.2.1.4 Frequent (≥ 1%) Adverse Events by Preferred Term in Decreasing Frequency

TEAEs occurring for at least 1% of the subjects in any of the treatment arms will be summarized by MedDRA PT in decreasing frequency of risankizumab treatment group.

### 9.2.1.5 Areas of Safety Interest

The Adverse Events of Safety Interest (ASI) categories will be summarized by SOC and PT and will be based on standardized or company MedDRA queries (SMQs or CMQs). Detailed information about the search criteria are provided in Appendix B. Adjudicated cardiovascular events will be summarized and presented by treatment group using the CAC adjudicated categories. Serious opportunistic infection excluding tuberculosis and herpes zoster, serious hypersensitivity, serious hepatic events and serious injection site reaction will also be summarized by PT. In addition, an overview of ASI per 100 patient-years of study exposure will be presented. The number of TEAEs reported, the total



number of years of study drug exposure, and the TEAE rate per 100 patient-years will be presented.

Similarly, overview tables for serious ASI in number and percentage as well as in event rate per 100 patient-years will be provided.

Additional AEs in ASI may be considered for tabulation/summary based on recommendations from Clinical and Safety teams, as deemed appropriate.

### 9.2.2 Analysis of Adverse Events for Long-Term

Long-term adverse event rates will be analyzed using event rates adjusted by cumulative exposure and will be based on the actual treatment received at the time of AE occurrence for the Any risankizumab 150 mg group. This includes AEs occurred under risankizumab 150 mg exposure from subjects starting on risankizumab 150 mg and subjects switching from placebo to risankizumab 150 mg.

## 9.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure

An overview of TEAE per 100 patient-years of study exposure will be presented for the AE categories defined in Section 9.2.1.1.

An overview of ASIs per 100 patient-years of study exposure will be presented similarly.

## 9.2.2.2 Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT

The TEAE rate per 100 patient-years of exposure will be calculated overall, for each SOC and PT, for the same AEs defined in Section 9.2.1 and reported for Any risankizumab 150 mg group.



## 9.2.2.3 Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation

SAEs (including deaths) and AEs leading to study drug discontinuation will be listed in tables, besides summary by SOC and PT covered in Section 9.2.2.2.

## 9.2.2.4 Areas of Safety Interest Rates per 100 Patient-Years of Study Drug Exposure

The ASI categories will be summarized and presented for the Any risankizamub 150 mg group using SOC and MedDRA PT. The ASI categories will be identified per Standard MedDRA Queries (SMQs)/Company MedDRA Queries (CMQs) in Appendix B. Serious opportunistic infection excluding tuberculosis and herpes zoster, serious hypersensitivity, serious hepatic events and serious injection site reaction will also be summarized by PT for the Any risankizamub 150 mg group.

The ASI rate per 100 patient-years of exposure will be calculated overall, for each SOC and each PT, for each of the category listed in Appendix B.

Similarly, overview table for serious ASI rate per 100 patient-years of exposure will be summarized.

### 9.3 Analysis of Laboratory Data

Data collected from central and local laboratories, including additional laboratory testing due to an SAE, will be used in all analyses, except for Baseline where SAE-related laboratory assessments on or before the first dose of study drug will be excluded. The clinical laboratory tests defined in the protocol operations manual (e.g., hematology and clinical chemistry) will be summarized.

Each laboratory variable will be summarized for all time points (starting with Baseline) with the number of non-missing observations, mean and standard deviation, median, minimum and maximum. Mean change from baseline to each applicable post-baseline visit will be summarized for selected laboratory variables to compare the treatment



difference between risankizumab 150 mg and placebo in Period 1. The number of observations, baseline mean, visit mean as well as the change from baseline mean, standard error, and 95% confidence interval within each treatment group and between treatment groups (risankizumab 150 mg vs. placebo) will be presented.

Changes in laboratory parameters will be tabulated using shift tables by CTCAE criteria v4.03 (Appendix H).<sup>1</sup> A shift table from baseline to the worse value (based on CTCAE criteria v4.03) during treatment will be created. A similar shift table will be provided to summarize shifts from baseline to the final post-baseline value.

Laboratory abnormalities meeting CTCAE criteria grade 3 and higher will be summarized.

Laboratory abnormalities will be evaluated based on Potentially Clinically Significant (PCS) criteria (Appendix C). For each laboratory PCS criterion, the number and percentage of subjects who have a laboratory value meeting the criteria will be summarized. Listings will be provided to summarize subject-level laboratory data for subjects meeting PCS criteria. A listing of possible Hy's Law cases will be provided.

#### 9.3.1 Variables and Units

All laboratory parameters to be collected in this study are listed below. Laboratory parameters will be reported using the standard international (SI) units.

Table 2. List of Laboratory Variables

| Laboratory Variables |
|------------------------------|
| Hematology |
| White Blood Cell (WBC) Count |
| Red Blood Cell (RBC) Count |
| Hemoglobin |
| Hematocrit |
| Platelets count |
| Neutrophils |



## Table 2. List of Laboratory Variables (Continued)

| Laboratory Variables Hematology (Continued) Basophils Eosinophils |
|----------------------------------------------------------------------|
| Basophils |
| Fosinophils |
| Losinopinis |
| Lymphocytes |
| Monocytes |
| Chemistry |
| Total Bilirubin |
| Alkaline Phosphatase (ALP) |
| Aspartate aminotransferase (AST) |
| Alanine aminotransferase (ALT) |
| Total Protein |
| Albumin |
| Glucose |
| Triglycerides |
| Blood Urea Nitrogen (BUN) |
| Creatinine |
| Sodium |
| Potassium |
| Calcium |
| Chloride |
| Bicarbonate |
| Gamma Glutamyl Transferase (GGT) |
| Cholesterol |
| LDL cholesterol |

## 9.3.2 Analysis of Laboratory Data for Period 1

HDL cholesterol

The laboratory data will be summarized by the actual treatment groups (risankizumab 150 mg and placebo group).



# 9.3.2.1 Assessment of Mean Change from Baseline in Clinical Laboratory Variables

Analyses of key continuous hematology and chemistry variables which are measured longitudinally will be performed by visits and by treatment group. For each parameter at each visit, the following summary statistics will be presented for each treatment group: sample size, mean, standard deviation, minimum, median and maximum.

An ANOVA model with treatment as a factor will be used to compare change from baseline between different treatment groups for selected laboratory parameters. Mean difference from placebo and associated 95% CIs will be presented. The analysis applies to the following laboratory parameters of clinical interest:

- Hematology parameters: WBC, neutrophils, lymphocytes, RBC, hematocrit, hemoglobin, platelets count.
- Chemistry parameters: total bilirubin, GGT, ALP, SGOT/AST, SGPT/ALT, glucose, creatinine, potassium, sodium, calcium.

## 9.3.2.2 Assessment of Shift from Baseline in Clinical Laboratory Variables

The baseline and post-baseline laboratory observations will be categorized as Grade 0, Grade 1, Grade 2, Grade 3, and Grade 4 and shifts from baseline grade to worst ontherapy grade will be summarized. A similar shift table will be provided to summarize shifts from baseline to the final post-baseline value. Toxicity grading scale is based on CTCAE version 4.03. Shift tables from baseline according to the grades will be provided for laboratory variables including SGPT/ALT, SGOT/AST, GGT, ALP, total bilirubin, creatinine, hemoglobin, neutrophils count, WBC, and lymphocyte count.

Note that the minimum/maximum category is used, rather than the category of the minimum/maximum value. The two may be different due to variation in the reference range.



No statistical tests will be performed for this analysis.

## 9.3.2.3 Assessment of Potentially Clinically Significant Laboratory Values

Laboratory abnormalities will be evaluated based on PCS criteria (Appendix B) (defined as a lab value  $\geq$  grade 3 NCI CTCAE v4.03 severity). For each laboratory PCS criterion, the number and percentage of subjects who have at least one post-baseline on-treatment value meeting the criteria will be summarized by actual treatment group. A listing of all observations collected will be generated for subjects who have at least one post-baseline observation meeting pre-defined criteria for potentially clinically significant values. A post baseline value must be more extreme than the baseline value to be considered a potentially clinically significant finding.

#### 9.3.2.4 Assessment of Liver Function Test Elevations

According to FDA's Guidance for Industry "Drug-Induced Liver Injury: Premarketing clinical evaluation" (July 2009), when aminotransferase abnormalities indicating hepatocellular injury are accompanied by evidence of impaired hepatic function (bilirubin elevation > 2 × ULN), in the absence of evidence of biliary obstruction (i.e., significant elevation of ALP) or some other explanation of the injury (e.g., viral hepatitis, alcohol hepatitis), the combined finding (i.e., Hy's Law cases) represents a signal of a potential for the drug to cause severe DILI.

For the purpose of assessing for potential Hy's law cases, the frequencies and percentages of subjects with post baseline liver specific function test values that meet the following criteria of potential clinical interest will be summarized by treatment groups:

- ALT  $\geq$  3 × ULN
- ALT  $\geq$  5 × ULN
- ALT  $\geq 10 \times ULN$
- ALT  $> 20 \times ULN$
- AST  $\geq$  3 × ULN



- $AST > 5 \times ULN$
- AST  $\geq 10 \times ULN$
- AST  $\geq 20 \times ULN$
- TBL  $\geq$  2 × ULN
- Alkaline phosphatase  $\geq 1.5 \times ULN$
- ALT and/or AST  $\geq$  3 × ULN and concurrent TBL  $\geq$  1.5 × ULN
- ALT and/or AST  $\geq$  3 × ULN and concurrent TBL  $\geq$  2 × ULN

A listing of potentially clinically significant liver function laboratory values will also be provided.

In addition, the Evaluation of Drug-Induced Serious Hepatotoxicity (eDISH) plot<sup>2</sup> will be generated to evaluate the liver safety profile of risankizumab. eDISH plot is a log/log display of correlation between peak total bilirubin (TBIL) vs. ALT, both in multiples of ULN, with horizontal and vertical lines indicating Hy's law thresholds, i.e.,  $ALT = 3 \times ULN$  and total bilirubin =  $2 \times ULN$ . The eDISH plot makes immediately evident subjects potentially matching Hy's law laboratory criteria, all located in the upper right quadrant of the graph. Data points in the lower right quadrant, i.e., exceeding  $3 \times ULN$  for ALT, but being below  $2 \times ULN$  for total bilirubin, suggest an increased risk for liver injury as well, if incidence is differing between active treatment and control groups, however, not to the same extent and with less specificity as compared to Hy's law.





Fig. 1 eDISH plot, TBIL [× ULN] vs. ALT [× ULN] on a log/log scale, treatment by panel, pooled active versus control. *ULN* upper limit of normal, *ALT* alanine aminotransferase, *TBIL* total bilirubin

Note: Merz 2014.<sup>2</sup>

## 9.3.3 Analysis of Long-Term Laboratory Data

# 9.3.3.1 Assessment of Mean Change from Baseline in Clinical Laboratory Variables

Analyses of specified continuous hematology and chemistry variables which are measured longitudinally will be performed by visits and by actual treatment group sequences as described in Section 9.1. For each parameter, the following summary statistics will be presented for each treatment group sequence: sample size, mean, standard deviation, minimum, median and maximum.



## 9.3.3.2 Assessment of Potentially Clinically Significant Laboratory Values

Long-term laboratory data will also be summarized based on the number and percentage of subjects meeting the criteria for potentially clinically significant (PCS) laboratory values for the Any Risankizumab 150 mg group.

The baseline value will be determined by the last non-missing measurement recorded on or before the date of the first dose of risankizumab 150 mg. For a subject who started on placebo and switched to risankizumab 150 mg at Week 24, lab values under risankizamab 150 mg exposure would be evaluated against the baseline value defined as above.

A listing of all subjects with any laboratory determination meeting CTCAE criteria of Grade 3 or higher will be provided by Grade. For each of these subjects, the whole course of the respective parameter will be listed.

#### 9.3.3.3 Assessment of Liver Elevations

The frequencies and percentages of subjects with post-baseline liver-specific function test values that meet the criteria of potential clinical interest defined in Section 9.3.2.4 will be summarized for Any risankizumab 150 mg group. A listing of potentially clinically significant liver function laboratory values will also be provided. For each of these subjects, the whole course of the respective parameter will be listed.

In addition, the eDISH plot as defined in Section 9.3.2.4 will be provided for Any risankizumab group.

## 9.4 Analysis of Vital Signs

Vital sign measurements of weight, systolic and diastolic blood pressure, and pulse rate will be summarized.

Vital sign variables will be evaluated based on potentially clinically significant (PCS) criteria (Appendix C).



### 9.4.1 Analysis of Vital Sign for Period 1

Analyses of continuous vital sign variables which are measured longitudinally will be performed by visits and by the treatment groups of risankizumab 150 mg and placebo group. For each analysis, the following summary statistics will be presented for each treatment group: sample size, mean, standard deviation, minimum, median and maximum.

The number and percentage of subjects meeting the criteria for PCS vital sign values will be summarized by actual treatment group. Listings will be provided to summarize subject-level vital sign data for subjects meeting PCS criteria. For each of these subjects, the whole course of the respective parameter will be listed.

### 9.4.2 Analysis of Long-Term Vital Sign

Analyses of continuous vital signs variables which are measured longitudinally will be performed by visits and by actual treatment group sequences as described in Section 9.1.

Long-Term vital sign will also be summarized based on the number and percentage of subjects meeting the criteria for PCS vital sign values for the Any risankizumab 150 mg group. A listing of all subjects with any vital sign values meeting the criteria for PCS vital signs will also be provided.

## 10.0 Other Analyses

No other analyses are planned.

## 11.0 Interim Analyses

Interim analyses may be conducted as deemed appropriate.

### 11.1 Data Monitoring Committee

An external independent data monitoring committee (DMC) will review unblinded safety data at regular intervals during the conduct of the study. The primary responsibility of the



DMC will be to protect the safety of the subjects participating in this study. When needed, high-level unblinded efficacy data may be requested by the DMC and be reviewed so that the DMC can assess benefit: risk of any emerging safety differences.

A separate DMC charter describes the roles and responsibilities of the DMC members, frequency of data reviews, relevant data to be assessed, and general operations.

## 12.0 Overall Type-I Error Control

A multiple testing procedure will be used to provide strong control of the type 1 error rate at alpha = 0.05 (2-sided) across analyses comparing risankizumab versus placebo with respect to the primary and the ranked secondary endpoints for Period 1.<sup>3</sup> Specifically, the testing will utilize a fix sequence of hypothesis testing for the primary endpoint followed by the ranked secondary endpoints in the order as specified in Section 3.2. The test starts with the primary endpoint using two-sided  $\alpha = 0.05$ ; testing can be conducted for a lower ranked endpoint only if the previous endpoints in the sequence meet the requirement of statistical significance.

The graph for the testing procedure is provided in Figure 3. In the graph, the arrows specify the  $\alpha$  transfer paths. Once an endpoint is rejected (i.e., deemed statistically significant) at its assigned significance level, its significance level will be transferred to the subsequent endpoint following the arrow.

Figure 3. Graphical Testing Procedure





## Figure 3. Graphical Testing Procedure (Continued)

ACR 20 = 20% improvement in American College of Rheumatology criteria; CFB = change from baseline; FACIT-Fatigue = Functional Assessment of Chronic Illness Therapy-Fatigue; HAQ-DI = Health Assessment Questionnaire-Disability Index; LDI = Leeds Dactylitis Index; LEI = Leeds Enthesitis Index; (PsA-) mTSS = Modified Total Sharp Score; MDA = minimal disease activity; PASI 90 = 90% improvement in Psoriasis Area and Severity Index in subjects with BSA  $\geq$  3% at Baseline; PGA-F = Physician's Global Assessment of Fingernails Psoriasis; mNAPSI = modified Nail Psoriasis Severity Index; SF-36 PCS = Short Form-36 Physical Component Summary

## 13.0 Version History

Table 3. SAP Version History Summary

| Version | Date | Summary |
|---|---|---|
| 1.0 | 04 Aug 2017 | Original version |
| 2.0 | 23 Aug 2018 | The following changes have occurred between the first version and the second version in order to reflect changes in the protocol and regulatory feedback. |
| | | <ul> <li>An update to the study design.</li> </ul> |
| | | <ul> <li>The addition of the Analysis Population And<br/>Important Subgroups section</li> </ul> |
| | | <ul> <li>The addition of the Demographics and<br/>Baseline Characteristics section</li> </ul> |
| | | • The addition of subgroups and modification from 2 to 3 categories for Baseline BMI. |
| | | • The addition of BASDAI 50 response to Section 7.0. |
| | | <ul> <li>Change in the order of the ranked secondary endpoints</li> </ul> |
| | | Addition of several non-ranked secondary endpoints |
| | | <ul> <li>Changes in the interim analysis section to<br/>reflect unblinded analyses</li> </ul> |
| | | <ul> <li>Changes in the missing data section to reflect<br/>changes in the planned analysis and<br/>sensitivity analyses</li> </ul> |
| | | <ul> <li>Changes in the safety analysis section in<br/>order to detail short and long term safety<br/>analyses.</li> </ul> |
| | | <ul> <li>Various editorial changes to enhance readability.</li> </ul> |



## Table 3. SAP Version History Summary (Continued)

| Version | Date | Summary |
|---|---|---|
| 3.0 | 25 Feb 2019 | The following changes have occurred between the second version and the third version in order to reflect changes in the protocol and regulatory feedback. |
| | | <ul> <li>An update to the study design to add bilateral radiographs to the Week 100 study visit.</li> <li>Remove references to US and ex-US subjects throughout the document as they relate to Secondary Endpoints assessing nail psoriasis (i.e., PGA-F vs. mNAPSI)</li> </ul> |
| | | Update Section 13.0 (Safety Analyses) to<br>reflect that Period 1 analyses will be<br>performed at Week 24 and Week 52. |
| 4.0 | 30 Mar 2020 | In addition to changes to adhere to a new SAP formatting standard the following additional sections have been included between the third version and the fourth version in order to add additional information. Subject Disposition Study Drug Duration and Compliance Medical History Prior and Concomitant Medications The following changes have occurred in order to reflect changes in the protocol and regulatory guideline. Updated secondary endpoints including replacing change from baseline in LDI/LEI with resolution of LDI/LEI as ranked secondary endpoints as well as adding ACR50/70 as other secondary endpoints. Added estimand language for primary and secondary endpoints. Provided analysis details for efficacy analysis in double-blind period and long-term efficacy analysis, including but not limit to, supplementary analysis for primary and secondary endpoints (e.g., MI, tipping point analysis), sensitivity analysis of primary endpoint based on Per Protocol analysis set. Revised multiple testing procedure by removing Hochberg. |
| | | Revised and provided analysis details for safety analysis including but not limit to ASI, lab mean change summary, PCS grading. |



 Table 3.
 SAP Version History Summary (Continued)

| Version | Date | Summary |
|---|---|---|
| 5.0 | 15 Sep 2020 | <ul> <li>The following changes have occurred</li> <li>Updated missing data handling due to COVID-19 infection or logistic restrictions</li> <li>Updated intercurrent event definition.</li> <li>Added ACR20 at Week 16 as ranked secondary endpoint.</li> <li>Updated resolution of LDI and resolution of LEI for subjects from pooled M15-998 and M16-011 data as ranked secondary endpoint</li> <li>Added additional efficacy endpoints related to BASDAI and ASDAS.</li> </ul> |
| | | Updated break-down summary of non-responders for<br>ACR20 at Week 24. |
| 6.0 | 23 Nov 2020 | <ul> <li>The following changes have occurred:</li> <li>Added rescue medication summary</li> <li>Updated tipping point analysis for mTSS using AO data and added MI using AO data</li> <li>Removed AE by relationship /severity in E/100PY in long-term</li> <li>Removed fungal infections and added serious anaphylactic reaction in ASI.</li> <li>Updated laboratory parameters of clinical interest for the treatment comparison</li> <li>Updated liver elevations criteria according to FDA's Guidance for Industry "Drug-Induced Liver Injury (July 2009)</li> </ul> |

## 14.0 References

- 1. National Cancer Institute. CTCAE v. 4.0. Available from: http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm#ctc.
- 2. Merz M, Lee KR, Kullak-Ublick GA, et al. Methodology to assess clinical liver safety data. Drug Saf. 2014;37 (Suppl 1):S33-45.
- 3. Bretz F, Maurer W, Brannath W, et al. A graphical approach to sequentially rejective multiple test procedures. Stat Med. 2009;28(4):586-604.



- 4. Greenland S, Rothman KJ. "Introduction to Stratified Analysis." In: Rothman KJ, Greenland S, Lash TL, editors. In Modern Epidemiology, 3<sup>rd</sup> ed. Philadelphia: Lippincott Williams & Wilkins; 2008. 258-82.
- 5. Rubin, DB. Multiple Imputation for Nonresponse in Surveys. New York: John Wiley & Sons Inc; 1987.
- 6. Carpenter JR, Kenward MG. Multiple Imputation and Its Application. New York: John Wiley & Sons; 2013.



## **Appendix A.** Protocol Deviations

The number and percentage of subjects who reported at least one of the following protocol deviation categories will be provided.

- Subject entered into the study even though s/he did not satisfy entry criteria.
- Subject developed withdrawal criteria during the study and was not withdrawn.
- Subject received wrong treatment or incorrect dose of study drug.
- Subject took prohibited concomitant medication.



## Appendix B. Definition of Areas of Safety Interest

The Adverse Events of Safety Interest (ASI) will be identified using the following search criteria:

| ASI | Search Criteria | |
|---|---|---|
| MACE | Adjudicated terms will be identified using CECAT and CETERM from the CE SDTM dataset. | |
| Extended MACE | | Adjudicated terms will be identified (for MACE +) using CECAT and CETERM from the CE SDTM dataset. |
| Serious Infections | Serious Al | Es in the Infections and Infestations SOC |
| Active Tuberculosis | Active Tul | berculosis CMQ (code 80000188) |
| Opportunistic Infection excluding tuberculosis and herpes zoster | | Opportunistic Infection excluding tuberculosis and herpes zoster CMQ (code 80000189) |
| Herpes Zoster | Herpes Zo | ster CMQ (code 80000175) |
| Malignant Tumours | Narrow | Malignant tumours (SMQ 20000194) |
| Non-melanoma Skin<br>Cancer (NMSC) | Broad Skin malignant tumours (SMQ 20000204) excluding terms identified b the Melanoma CMQ (code 80000119) | |
| Malignant Tumours excluding NMSC | 'Malignant Tumours excluding NMSC' is identified by the 'Malignant Tumours' search excluding terms identified by the 'Non-melanoma skin cancer (NMSC)' search. | |
| Hypersensitivity | Narrow | Narrow Hypersensitivity (SMQ 20000214) |
| Serious Anaphylactic<br>Reactions | Narrow Serious AEs in the Anaphylactic Reaction SMQ (SMQ 20000021) | |
| Adjudicated Anaphylactic Reactions* | Adjudicate | ed terms will be identified using SDTM data (e.g., CE and PR domains). |
| Hepatic Events | Broad | Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions (SMQ 20000013) |
| | Broad | Hepatitis, non-infectious (SMQ 20000010) |
| | Broad | Cholestasis and jaundice of hepatic origin (SMQ 20000009) |
| | Broad | Liver related investigations, signs and symptoms (SMQ 20000008) |
| | Narrow | Liver-related coagulation and bleeding disturbances (SMQ 20000015) |
| Injection Site Reactions | Injection S | Injection Site Reaction CMQ (code 80000019) |

<sup>\*</sup> Events will be identified for adjudication by Anaphylactic Reaction SMQ Broad search as specified in the RISA AAC Charter.

## Appendix C. Potentially Clinically Significant Criteria for Safety Endpoints

The criteria for Potentially Clinically Significant (PCS) laboratory findings are described in Table C-1 and Table C-2, and the PCS criteria for vital sign findings are described in Table C-3.

Table C-1. Criteria for Potentially Clinically Significant Hematology Values

| | | Definition of Potentially Clinically Significant<br>Current (Version 4) CTCAE Grade 3 or Greater |
|---|---|---|
| Hematology Variables | Units | Very Low |
| Hemoglobin | g/dL | < 8.0 |
| Platelets count | 10 <sup>9</sup> /L | < 50.0 |
| WBC count | 10 <sup>9</sup> /L | < 2.0 |
| Neutrophils | 10 <sup>9</sup> /L | < 1.0 |
| Lymphocytes | 10 <sup>9</sup> /L | < 0.5 |

Table C-2. Criteria for Potentially Clinically Significant Chemistry Values

| | | Definition of Potentially Clinically Significant Current<br>(Version 4) NCI CTCAE Grade 3 or Greater | |
|---|---|---|---|
| <b>Chemistry Variables</b> | Units | Very Low | Very High |
| TBL | mcmol/L | | > 3.0 × ULN |
| ALP | U/L | | $> 5.0 \times \text{ULN}$ |
| SGOT/AST | U/L | | $> 5.0 \times \text{ULN}$ |
| SGPT/ALT | U/L | $> 5.0 \times ULN$ | |
| Albumin | g/L | < 20 | |
| Glucose | mmol/L | < 2.2 | > 13.9 |
| Creatinine | mcmol/L | | $> 3.0 \times ULN (> 3.0 \times BL)$ |
| Sodium | mmol/L | < 130 | > 155 |
| Potassium | mmol/L | < 3.0 | > 6.0 |
| Calcium | mmol/L | < 1.75 | > 3.1 |
| GGT | | | > 5.0 × ULN |



## Table C-3. Criteria for Potentially Clinically Significant Vital Sign Values

| Vital Sign | Category | Criteria for Potential Clinically Significant Vital Signs |
|---|---|---|
| Systolic blood pressure | Low | Value ≤ 90 mmHg and decrease ≥ 20 mmHg from Baseline |
| | High | Value $\geq 160$ mmHg and increase $\geq 20$ mmHg from Baseline |
| Diastolic blood pressure | l pressure Low Value ≤ 50 mmHg and decrease ≥ 10 mmH | |
| | High | Value ≥ 100 mmHg and increase ≥ 10 mmHg from Baseline |



# Appendix D. Definition of Estimand for Primary and Ranked Secondary Endpoints

| | Attributes of the Estimand | | | | |
|---|---|---|---|---|---|
| Estimand | Treatments | Population | Variable | Intercurrent<br>Events (IE) | Population<br>Level<br>Summary |
| Composite estimand for binary endpoints <sup>a</sup> (primary) | Risakizumab<br>150 mg vs<br>placebo | Subjects who randomized and received at least one dose of study drug. | ACR20/50/ 70 response/ PASI90 response/MDA response/ resolution of LEI/resolution of LDI at Week 24 and ACR 20 at Week 16 (initiation of concomitant medications for PsA that could meaningfully impact efficacy assessment or rescue as non- responder) | The IE is captured through the variable definition | Difference in response proportions between treatment conditions |
| Treatment policy estimand for binary endpoints <sup>a</sup> (supplementary) | Risakizumab 150 mg vs placebo (regardless of adherence to study drug or initiation of concomitant medications for PsA that could meaningfully impact efficacy assessment or use of rescue medication) | Subjects who randomized and received at least one dose of study drug. | ACR20/50/70 response/ PASI90 response/MDA response/ resolution of LEI/resolution of LDI at Week 24 and ACR20 at Week 16 | The IE is captured through the treatment definition | Difference<br>in response<br>proportions<br>between<br>treatment<br>conditions |



| | Attributes of the Estimand | | | | |
|---|---|---|---|---|---|
| Estimand | Treatments | Population | Variable | Intercurrent<br>Events (IE) | Population<br>Level<br>Summary |
| Hypothetical estimand for continuous endpoints <sup>b</sup> (primary) | Risakizumab<br>150 mg vs<br>placebo | Subjects who randomized and received at least one dose of study drug. | Change from<br>baseline in<br>HAQ-DI<br>/mNAPSI /<br>PGA-F/SF-36<br>(PCS)/FACIT-<br>fatigue at<br>Week 24 | Had subjects not started initiation of concomitant medications for PsA that could meaningfully impact efficacy assessment or not rescued | Difference<br>in variable<br>means<br>between<br>treatment<br>conditions |
| Hypothetical estimand for continuous radiographic endpoint <sup>c</sup> (primary) | Risakizumab<br>150 mg vs<br>placebo | Subjects who randomized and received at least one dose of study drug. | Change from baseline in mTSS | Had subjects<br>not<br>prematurely<br>discontinued<br>study drug or<br>not rescued | Difference<br>in variable<br>means<br>between<br>treatment<br>conditions |
| Treatment policy estimand for continuous endpoints <sup>b</sup> and continuous radiographic endpoint <sup>c</sup> (supplementary) | Risakizumab 150 mg vs placebo (regardless of concomitant medications use for PsA that could meaningfully impact efficacy or adherence to study drug or use of rescue medication) | Subjects who randomized and received at least one dose of study drug. | Change from<br>baseline in<br>HAQ-DI/mTSS<br>/mNAPSI/<br>PGF-F/SF-36<br>(PCS)/FACIT-<br>Fatigue at Week<br>24 | The IE is captured through the treatment definition | Difference<br>in variable<br>means<br>between<br>treatment<br>conditions |

- a. Binary endpoints include ACR20/50/70, PASI90, MDA, resolution of LEI and resolution of LDI.
- b. Continuous endpoints include HAQ-DI, mNAPSI, PGA-F, SF-36 (PCS), FACIT-fatigue.
- c. Continuous radiographic endpoint includes mTSS.

#### **Appendix E.** NRI-C Procedure

### **Composite Binary Endpoints**

### Step 1:

Missing binary values are first imputed via MI under MAR assumption using the FCS method with the logistic regression option. The FCS method can handle any arbitrary missing data pattern, without monotone missing requirement. Treatment is included in the FCS imputation model to enable stratified sampling conditional on treatment groups. The imputation model includes gender, race (white vs. non-white), ethnicity, age, baseline BMI, geographic regions, duration of PsA, baseline values of the components of the composite binary endpoint, stratification factors, intercurrent event status, as well as longitudinal response observed at any other visits. The number of imputed datasets is 30 for each PROC MI. Sample codes are as follows:

```
proc mi data=data2 seed=&seed nimpute=30 out=mar_imp;
class &predcate &postout;
fcs logistic;
by treatment;
var &predcate &predcont &postout;
run;

&predcate (categorical covariates): gender, race (white vs. non-white),
ethnicity, geographic regions, concomitant csDMARD at baseline(yes vs
no), extent of psoriasis, presence of dactylitis, presence of enthesitis
and intercurrent event status. &predcont (continuous covariates): age,
baseline BMI, duration of PsA, baseline components. &postout: Binary
endpoint at week 4, 8, 12, 16, 24
```

#### Step 2:

For each imputed dataset, the imputed response status for missing due to reasons other than COVID-19 is overridden by NRI to ensure that multiple imputation is only applied to missing due to COVID-19. Subjects will be considered as non-responders after initiation of rescue medication or initiation of concomitant medications for PsA that could



meaningfully impact efficacy assessment (including COVID-19 impacted visits of which response status is imputed by MI in step 1).

#### Step 3:

For each of the 'complete' datasets, the CMH test is performed adjusting the stratification factors to estimate the treatment difference of risankizumab versus placebo and the corresponding standard error. The SAS procedure PROC STDRATE is used to compute the treatment difference, corresponding 95% CI and p-value adjusting for stratification factors using the Mantel-Haenszel method (Greenland and Rothman 2008, p. 271).<sup>4</sup> Sample SAS codes are as follows:

```
proc stdrate data=data2 method=mh stat=risk effect=diff;
population group=TRTP event=N_RESPONDERS total=N_TOTAL;
strata STRATA / order=data stats effect;
run:
```

Note: The input dataset is summary level data including the following variables: treatment group (denoted by TRTP), stratification factors (denoted by STRATA), number of responders per study and treatment group (denoted by N RESPONDERS) and total number of subjects per study and treatment group (denoted by N TOTAL).

The results from the 30 'complete' datasets will be synthesized using the SAS procedure PROC MIANALYZE, following Rubin's formula (Rubin, 19874)<sup>5</sup>, to derive the MI estimator of the treatment difference for the final statistical inferences. Sample SAS codes are as follows:

```
proc mianalyze data=data3;
modeleffects RiskDiff;
stderr StdErr;
ods output parameterestimates=risk_diff_mh;
run;
```



#### **Binary Endpoints Dichotomized from Continuous Scale**

#### Step 1:

When a dichotomized variable is derived from a continuous scale, the MI is applied to the original continuous scale. Missing values are imputed via MI with the FCS method. Treatment is included in the FCS imputation model to enable stratified sampling conditional on treatment groups. The imputation model includes gender, race (white vs. non-white), ethnicity, age, baseline BMI, geographic regions, duration of PsA, baseline value of the endpoint of interest (in continuous scale), stratification factors, intercurrent event status, as well as longitudinal response (in continuous scale) observed at any other visits. The number of imputed datasets is 30 for each PROC MI. Sample codes are as follows:

```
proc mi data=data1 seed=&seed nimpute=30 out=mar_imp; class &predcate; fcs; by treatment; var &predcate &predcont &postout; run;

Note: &predcate (categorical covariates): gender, race (white vs. non-white), ethnicity, geographic regions, concomitant csDMARD at baseline (yes vs no), extent of psoriasis, presence of dactylitis, presence of enthesitis and intercurrent event status. &predcont (continuous covariates): age, baseline BMI, duration of PsA, baseline value. &postout: continuous scale of the binary endpoint at week 4, 8, 12, 16, 24
```

The dichotomized variable is then derived from the imputed value for each imputed dataset.

#### Step 2:

For each imputed dataset, the imputed response status for missing due to reasons other than COVID-19 is overridden by NRI to ensure that multiple imputation is only applied to missing due to COVID-19. Subjects will be considered as non-responders after initiation of rescue medication or initiation of concomitant medications for PsA that could



meaningfully impact efficacy assessment, including COVID-19 impacted visits of which response status is imputed by MI in step 1.

### Step 3:

For each of the 'complete' datasets, the CMH test is performed adjusting the stratification factors to estimate the treatment difference of risankizumab versus placebo and the corresponding standard error. The results from the 30 'complete' datasets will be synthesized using the SAS procedure PROC MIANALYZE, following Rubin's formula (Rubin, 19874)<sup>5</sup>, to derive the MI estimator of the treatment difference for the final statistical inferences. Sample codes follow the same as provided above for composite binary endpoints (step 3).

### Appendix F. Tipping Point Analysis for Non-Radiographic Endpoints

#### **Tipping Point Analysis for ACR20**

To assess the robustness of the primary analysis using NRI-C data handling, tipping point analysis is conducted on ACR20 at Week 24.

The analysis is conducted on the FAS using AO data, i.e., all observed data regardless of concomitant medications use for PsA, study drug adherence or rescue.

The tipping point analyses are two-dimensional, i.e., assumptions about the missing outcomes on the risankizumab treatment group and the placebo group can vary independently. Missing binary values are first imputed via MI under MAR assumption using the FCS method with the logistic regression option.

Two sets of shift parameters are applied to the imputed values by adding two MNAR statements to the same PROC MI, which allow the missing response rate to systematically vary from 0% to 100% in both risankizumab and placebo, respectively. This is accomplished by modifying the predicted probabilities for the responses through shifting the log odds (shift parameters are log odds ratios)<sup>6</sup>, then directly sampling the missing response from the Bernoulli distribution with the modified probabilities. Sample codes are as follows:

```
proc mi data=data2 seed=&seed nimpute=30 out=mnar_imp;
class &predcate &postout;
fcs reg(BLj= &predcate &predcont, excluding BL);
fcs logistic(week4=&predcate &predcont);
fcs logistic(week8=&predcate &predcont week4);
fcs logistic(week12=&predcate &predcont week4 week8)
fcs logistic(week12=&predcate &predcont week4 week8 week12);
fcs logistic(week24=&predcate &predcont week4 week8 week12);
by treatment;
var &predcate &predcont &postout;
mnar adjust(wk24(event="1") /shift=&sj1 adjustobs=(&treatment="PBO"));
mnar adjust(wk24(event="1") / shift=&sj2 adjustobs=(&treatment="RIS"));
run;

&predcate (categorical covariates): gender, race (white vs. non-white),
ethnicity, geographic regions, concomitant csDMARD at baseline (yes vs.)
```



no), extent of psoriasis, presence of dactylitis, presence of enthesitis, and intercurrent event status. &predcont (continuous covariates): age, baseline BMI, duration of PsA, 7 baseline ACR components. &postout: ACR20 binary values at week 4, week 8, week 12, week 16, week 24. BL $_{\rm J}$  is the jth baseline ACR components in the order of TJC, SJC, Pain, PGA, PhGA, HAQ-DI, CRP.

For each pair of shift parameters, the same CMH method used for the primary analysis will be performed on each of the multiple imputed datasets to obtain the results for each comparison of the risankizumab treatment group versus the placebo group adjusted by stratification factors. PROC MIANALYZE will then be used to aggregate the results for the final statistical inference using Rubin's method.

If one pair of shift parameters are found to just reverse the study conclusion, in terms of p-value larger than 0.05, then the shift parameters are identified as the tipping point. The results for a grid of shift parameter combinations are provided in tabular format.

### **Tipping Point Analysis for HAQ-DI**

To assess the impact of potential departures from the MAR assumption, tipping point analyses are conducted as a sensitivity check for change from baseline in HAQ-DI at Week 24.

The tipping point analyses are two-dimensional, i.e., assumptions about the missing outcomes on the risankizumab treatment groups and the placebo group can vary independently. Missing values are first imputed via MI under MAR using AO data, and then a shift parameter is applied to the imputed values (a different shift parameter may be specified for each treatment group). This is implemented by PROC MI using the MNAR statement. The imputation model uses FCS method, thus does not rely on a monotone missing pattern. It includes the same variables as for binary endpoint and is also stratified by treatment group. The number of imputed datasets is 30 for each PROC MI.

In cases where the shifted values are smaller than the minimum or larger than maximum value of the endpoint, (i.e., out of range), the minimum or maximum value of the endpoint is used in further analysis steps. For each pair of shift parameters, the SAS procedure



PROC MIXED is used for ANCOVA analysis which includes the fixed effects of treatment, the stratification factors and the continuous fixed covariate of baseline measurement on each of the imputed datasets to obtain the results for risankizumab treatment group versus the placebo group comparison. These results will be aggregated using Rubin's method to get p-values.

If one pair of shift parameters are found to just reverse the study conclusion, in terms of p-value larger than 0.05, then the shift parameters are identified as the tipping point. The results for a grid of shift parameter combinations are provided in tabular format.

## **Appendix G.** Details of Supplementary Analyses for Radiographic Continuous Endpoints

#### MI Analysis for Radiographic Continuous Endpoints

The MI analysis will impute missing data multiple times under appropriate random variation and thus generate multiple imputed "pseudo-complete" datasets. The imputation assumes of missing at random (MAR). ANCOVA will be performed on each of the multiple imputed datasets. The results will be aggregated across the multiple imputed datasets using Rubin's method. The SAS procedure PROC MI with the monotone statement and REGRESSION method is used. Before applying PROC MI, MCMC is applied where necessary to augment data into monotone missing pattern. The SAS code example for PROC MI is as follows:

```
PROC MI DATA=DATA WIDE1 OUT=DATA WIDE2 NIMPUTE=1 SEED=12345;
      Mcmc impute = monotone;
      VAR &COVCON WEEK 24;
       By trtp;
RUN:
PROC MI DATA=DATA WIDE2 OUT=OUTMI NIMPUTE=30 SEED=12345;
      CLASS &COVCAT;
      MONOTONE;
      VAR &COVCAT &COVCON WEEK 24;
       By trtp;
RUN;
Note:
       The input dataset is in wide format. TRTP denotes the treatment group. &COVCON denotes baseline
       continuous covariates including baseline age, baseline BMI, duration of PsA diagnosis and baseline value of
        the endpoint of interest. &COVCAT denotes categorical covariates including gender, race, ethnicity, regions,
        concomitant csDMARD at baseline (yes vs no), extent of psoriasis, presence of dactylitis, presence of
       enthesitis,. WEEK 24 denote the observed values at each visit.
PROC MIXED DATA=ALL;
     ODS OUTPUT LSMEANS=MIXEDLSMEANS DIFFS=DIFF;
     BY IMPUTATION ;
     CLASS TRTP STRATA;
```

```
MODEL CHG = BASELINE TRTP STRATA / SOLUTION;
    LSMEANS TRTP / CL PDIFF DIFF;
RUN;
DATA DIFF1;
    SET DIFF;
    COMPARISON= TRTP||' VS '||LEFT( TRTP);
RUN:
PROC SORT DATA=DIFF1; BY COMPARISON IMPUTATION ; RUN;
PROC MIANALYZE DATA=MIXEDLSMEANS1;
ODS OUTPUT PARAMETERESTIMATES=GROUP OUTPUT;
MODELEFFECTS ESTIMATE;
STDERR STDERR;
RUN;
PROC MIANALYZE DATA=DIFF1;
    ODS OUTPUT PARAMETERESTIMATES=GROUP OUTPUT;
    BY comparison;
   MODELEFFECTS ESTIMATE;
    STDERR STDERR;
RUN;
```

Note: The input dataset ALL includes all 30 imputed datasets. TRTP denotes the treatment group and STRATA denotes the stratification factor used in analysis. CHG denotes the change from baseline value and BASELINE denotes the baseline value.

#### **Tipping Point Analysis for Radiographic Continuous Endpoints**

To assess the impact of potential departures from the missing-at-random assumption, tipping point analyses are conducted as a sensitivity check for change from baseline in mTSS at the protocol defined primary time point.

The tipping point analyses are two-dimensional, i.e., assumptions about the missing outcomes on the risankizumab treatment groups and the placebo group can vary independently. In addition, the focus is on scenarios where missing outcomes on risankizumab are worse than the imputed values on risankizumab, while missing outcomes on placebo are better than the imputed values on placebo. Missing values are first imputed via MI under MAR, and then a shift parameter is applied to the imputed

Note:

values (a different shift parameter may be specified for each treatment group). This is implemented by PROC MI using the MNAR statement.

More specifically, PROC MI with the monotone statement and REGRESSION method will be performed to impute any missing value. Before applying PROC MI, MCMC is applied where necessary to augment data into monotone missing pattern. The number of imputed datasets is 30 for each PROC MI. Sample codes are as follows:

The input dataset is in wide format. TRTP denotes the treatment group. &COVCON denotes baseline continuous covariates including baseline age, baseline BMI, duration of PsA diagnosis and baseline value of the endpoint of interest. &COVCAT denotes categorical covariates including gender, race, ethnicity, regions, concomitant csDMARD at baseline (yes vs no), extent of psoriasis, presence of dactylitis and presence of enthesitis. WEEK 24 denote the observed values at each visit.

In cases where the shifted values are smaller than the minimum or larger than maximum value of the endpoint, (i.e., out of range), the minimum or maximum value of the endpoint is used in further analysis steps. For each pair of shift parameters, the SAS procedure PROC MIXED is used for ANCOVA analysis which includes the fixed effects of treatment, the stratification factors and the continuous fixed covariate of baseline measurement on each of the multiple imputed datasets to obtain the results for risankizumab treatment group versus the placebo group comparison. These results will be aggregated using Rubin's method to get p-values.



If one pair of shift parameters are found to just reverse the study conclusion, in terms of p-value larger than 0.05, then the shift parameters are identified as the tipping point. The results for a grid of shift parameter combinations are provided in tabular format.



## Appendix H. CTCAE Grades

| Test | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| SGPT/ALT increased | $>$ ULN $-3.0 \times$ ULN | $> 3.0 - 5.0 \times ULN$ | $> 5.0-20.0 \times ULN$ | $> 20.0 \times ULN$ |
| SGOT/AST increased | $>$ ULN $-3.0 \times$ ULN | $> 3.0 - 5.0 \times ULN$ | $> 5.0-20.0 \times ULN$ | $>20.0\times ULN$ |
| GGT increased | $>$ ULN $-2.5 \times$ ULN | $> 2.5 - 5.0 \times ULN$ | $> 5.0-20.0 \times ULN$ | $>20.0\times ULN$ |
| ALP increased | $>$ ULN $-2.5 \times$ ULN | $> 2.5 - 5.0 \times ULN$ | $> 5.0-20.0 \times ULN$ | $>20.0\times ULN$ |
| TBL increased | $>$ ULN $-1.5 \times$ ULN | $> 1.5 - 3.0 \times ULN$ | $>3.0-10.0\times ULN$ | $> 10.0 \times ULN$ |
| Creatinine <sup>†</sup> increased | >1 - 1.5 x baseline | >1.5 - 3.0 x BL; | >3.0 x BL; | $> 6.0 \times ULN$ |
| | (BL); > ULN –<br>1.5 × ULN | $> 1.5 - 3.0 \times ULN$ | $> 3.0 - 6.0 \times ULN$ | |
| Hemoglobin decreased* | < LLN - 100.0 g/L | < 100.0 - 80.0 g/L | < 80.0 - 65.0 g/L | < 65.0 g/L |
| Neutrophil count decreased | $< LLN - 1.5 \times 10^9/L$ | $< 1.5 - 1.0 \times 10^9 / L$ | $< 1.0 - 0.5 \times 10^9 / L$ | $<0.5\times10^9/L$ |
| WBC decreased | $\leq LLN - 3.0 \times 10^9/L$ | $< 3.0 - 2.0 \times 10^9/L$ | $< 2.0 - 1.0 \times 10^9 / L$ | $<1.0\times10^9/L$ |
| Lymphocyte count decreased | $< LLN - 0.8 \times 10^9/L$ | $< 0.8 - 0.5 \times 10^9 / L$ | $< 0.5 - 0.2 \times 10^9 / L$ | $< 0.2 \times 10^9 / L$ |

<sup>†</sup> If the calculation based on BL results in a different grade than the calculation based on ULN, use the higher grade.

<sup>\*</sup> Hemoglobin Grade 3 and Grade 4 are modified from CTCAE v4.



## Appendix I. Geographic Region

The following table lists the countries considered for each geographic region.

| Geographic Region | Countries |
|---|---|
| Asia | Malaysia, Singapore, South Korea, Taiwan, Israel |
| Eastern Europe | Bosnia and Herzegovina, Bulgaria, Croatia, Czech Republic, Estonia,<br>Hungary, Latvia, Lithuania, Poland, Romania, Russia, Serbia, Slovakia,<br>Ukraine |
| South/Central America | Argentina, Brazil, Chile, Mexico |
| North America | Canada, United States, Puerto Rico |
| Other | South Africa, Australia, New Zealand |
| Western Europe | Belgium, France, Germany, Greece, Ireland, Italy, Netherlands, Portugal, Spain, United Kingdom, Denmark, Finland, Sweden |